CLINICAL TRIAL: NCT03263858
Title: Vascular Implant Safety and Efficacy Study
Acronym: BIOVITESSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik CRC Inc. (Industry)
Collaborators: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1606
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Intervention Model Description: consecutive enrolment of cohort 1 (primary endpoint at 1 month), and cohort 2 (primary endpoint at 9 months)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 and 2 (Experimental)
  Interventions: Device: Stent

INTERVENTIONS:
Device: Stent — Implantation of coronary stent in de novo coronary artery lesions

SUMMARY:
Assessment of the safety and clinical performance of a coronary stent system in de novo coronary artery lesions

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years and < 85 years old
2. Written subject informed consent
3. Subjects with stable or unstable angina pectoris or documented silent ischemia or hemodynamically stable NSTEMI patients
4. Subject is eligible for percutaneous coronary intervention (PCI)
5. Subject is acceptable candidate for coronary artery bypass surgery
6. Subject is eligible for Dual Anti Platelet Therapy (DAPT)
7. Subjects with a maximum of two single discrete de novo lesions in two separate native coronary arteries that can be treated with the study stent during the index procedure
8. Reference vessel diameter of 3.0 mm to 3.8 mm by visual estimation.
9. Target lesion length up to 22 mm by visual estimation.
10. Target lesion with ≥ 50% and < 100% stenosis by visual estimation

Exclusion Criteria:

1. Left main coronary artery disease
2. Three-vessel coronary artery disease at the time of index procedure
3. Angiographic evidence of thrombus in target vessel
4. Chronic total occlusion
5. Heavily calcified or extremely tortuous lesions that would prevent complete inflation of a pre-dilatation balloon
6. Bifurcation lesion requiring side branch intervention, if side branches > 2mm in diameter are involved
7. Ostial lesions (within 5 mm of vessel origin)
8. In-stent restenosis
9. Lesions with prior treatment with a drug coated balloon (DCB)
10. Target lesion is located in or supplied by an arterial or venous bypass graft
11. Target lesion requires treatment with. rotational atherectomy
12. Proximal or distal to the target lesion located stenosis that might require future revascularization or impede run off detected during diagnostic angiography
13. Previous treatment of target vessel within 9 months of index-procedure
14. Patients with cardiogenic shock
15. Documented left ventricular ejection fraction (LVEF) ≤ 30%
16. Impaired renal function (serum creatinine > 2.5 mg/dl or 221 mmol/l, determined within 72 hours prior to intervention)
17. Hemodynamically unstable NSTEMI or STEMI within 72 hours prior to index procedure
18. Cerebrovascular event (within 3 months of index procedure)
19. Subject is receiving oral or intravenous immuno-suppressive therapy (inhaled steroids are allowed) or has known life-limiting immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus, but not diabetes mellitus)
20. Known allergies to: Acetylsalicylic Acid (ASA), heparin, contrast medium, sirolimus, or similar drugs, exipients or the stent material
21. Triple anticoagulation therapy
22. Life expectancy less than 1 year
23. Pregnant or breast-feeding females or females who intend to become pregnant during the time of the study
24. Inability to understand or read the informed consent form
25. Subject is currently participating in another study with an investigational device or an investigational drug and has not reached the primary endpoint yet
26. In the investigators opinion subjects will not be able to comply with the follow-up requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Strut coverage cohort 1 | 1 month
  Strut coverage will be assessed by OCT analysis
In stent late lumen loss cohort 2 | 9 months
  Late lumen loss with will be assessed by central QCA assessment

CONTACTS AND LOCATIONS:
Locations (5):
- Switzerland (5):
  - University Hospital Bern, Bern
  - Hôpiteaux Universitaires Genève (HUG), Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Cardiocentro Ticino, Lugano
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No